CLINICAL TRIAL: NCT03750890
Title: A New Strategy for the Visulation of Molecular Genotype in Glioma Evolution Based on the Radiomics and Microomics
Brief Title: Visual Study of Molecular Genotype in Glioma Evolution
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZWZ2018
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-11

CONDITIONS: Glioma of Brain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The key molecular changes in the progression of glioma are closely related to tumor heterogeneity, pathological grade, precision treatment and prognosis of glioma. At present, a visually quantitative assessment criteria about the key molecular typing of glioma is still absent. Based on the previous research, this project intends to establish a multi-dimensional database of glioma from clinical, radiomics and microomics levels. The investigators aim to filter out the specific molecular markers in the progression of glioma and explore the intrinsic connection of radiomics features and microomics molecular markers by using bioinformatics integration analysis and artificial intelligence multiple kernel learning. Thus, the investigators could determine the specific molecular mechanism in the progression of glioma, and establish a visually quantitative assessment system of pre-operative precisive grading, molecular typing discrimination and prognosis prediction. The completion of this project is of great significance for improving molecular diagnostic level of glioma, guiding individualized diagnosis and treatment decisions, and improving the survival rate of patients.

ELIGIBILITY:
Inclusion Criteria:

1. postoperative pathological and genetic test confirmed brain glioma;
2. The preoperative Clear and complete multimodal imaging data were collected within 10 days.

Exclusion Criteria:

1. patients who underwent surgery more than 4 weeks after MRI;
2. patients with motion artifacts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients who were suspected of having brain gliomas on the basis of clinical findings and who were previously diagnosed with brain gliomas underwent MRI.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
radiomics features（the parameters of T1WI, T2WI, DWI, DKI, ASL, ESWAN, DCE, MRS and so on） | through study completion, an average of 3 years
  the radiomics features（the parameters of T1WI, T2WI, DWI, DKI, ASL, ESWAN, DCE, MRS and so on）in the progression of glioma
microomics molecular markers (IDH mutation, 1p/19q status, P53 mutation, TERT and ATRX mutation, EGFR amplification and mutation, MGMT methylation status, PTEN mutation, ZM fusion gene and other gene features) | through study completion, an average of 3 years
  the key molecular markers (IDH mutation, 1p/19q status, P53 mutation, TERT and ATRX mutation, EGFR amplification and mutation, MGMT methylation status, PTEN mutation, ZM fusion gene and other gene features) in the progression of glioma

CONTACTS AND LOCATIONS:
Locations (1):
- Zhenxiong Wang, Wuhan, Choose A State Or Province, China